CLINICAL TRIAL: NCT02743715
Title: Randomized, Sham-Controlled Trial of Transcranial Direct Current Stimulation (tDCS) for Treatment-Resistant Obsessive-Compulsive Disorder (FRONT)
Brief Title: Transcranial Direct Current Stimulation (tDCS) for Treatment-Resistant Obsessive-Compulsive Disorder (FRONT)
Acronym: FRONT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Roseli Gedanke Shavitt, MD, PhD Department & Institute of Psychiatry Obsessive-Compulsive Spectrum Disorders Program University of Sao Paulo Medical School, Brazil, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FRONT2016
Record Dates: First submitted 2016-04-07; First posted 2016-04-19 (Estimated); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive-Compulsive Disorder; Transcranial direct current stimulation; Neuromodulation
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: randomized, sham-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: all study staff were blind to the participant's condition; only the neuromodulation staff, external to the study team, were aware of the participant's treatment group
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active tDCS (Active Comparator): Electric current of 2mA delivered to the cathode, positioned bilaterally in the cranial region corresponding to the supplementary motor cortex, with the anode positioned in the deltoid (neutral region), in 30-minute sessions, 5 days a week (Mondays through Fridays) for four consecutive weeks.
  Interventions: Device: Active tDCS (transcranial direct current stimulation)
- Sham tDCS (Sham Comparator): In this group, the cathode is positioned bilaterally in the cranial region corresponding to the supplementary motor cortex, with the anode positioned in the deltoid (neutral region), in 30-minute sessions, 5 days a week (Mondays through Fridays) for four consecutive weeks, without delivery of the electric current.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS (transcranial direct current stimulation) — An electrical current of 2mA is delivered to the cathode, positioned bilaterally in the cranial region corresponding to the supplementary motor cortex, with the anode positioned in the deltoid (neutral region), in 30-minute sessions, 5 days a week (Mondays through Fridays) for four consecutive weeks.
  Arms: Active tDCS
Device: Sham tDCS — The cathode is positioned bilaterally in the cranial region corresponding to the supplementary motor cortex, with the anode positioned in the deltoid (neutral region), in a 30-minute session, 5 days a week (Mondays through Fridays) for four consecutive weeks, without delivery of the electric current.
  Arms: Sham tDCS

SUMMARY:
Neuromodulation techniques for the treatment of Obsessive-Compulsive Disorder (OCD) have expanded with the greater understanding of the brain circuits involved in this disorder. Transcranial direct current stimulation (tDCS) is a non-invasive neuromodulation technique that has been studied as an alternative for strategy for treatment-resistant OCD. The main study is a randomized, sham-controlled, double-blinded trial tDCS for OCD patients unresponsive to cognitive-behavioral therapy and/or selective serotonin reuptake inhibitors. Forty-four patients will be randomized to two groups: active or simulated intervention. The intervention consisted of delivering an electric current of 2mA to the cathode, positioned bilaterally in the cranial region corresponding to the supplementary motor cortex, and the anode positioned in the deltoid (neutral region), during 30-minutes, for four consecutive weeks. The primary outcome was the reduction in baseline YBOCS scores before and after of tDCS treatment. Secondary outcomes include measures of depressive and anxiety symptoms, genetic markers, motor cortical excitability and performance in neurocognitive tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with OCD according to DSM IV criteria
* YBOCS score of 16 and above or ≥10 (for the presence of only compulsions or only obsessions)
* Patients with other psychiatric comorbidities are not excluded, however, OCD should be the most important disease .
* Age between 18 and 65
* Patients who failed one or more treatments
* Patients with no previous treatment for OCD will be treated with one first line treatment before being considered to participate in the tDCS trial.
* Voluntary and competent to consent

Exclusion Criteria:

* Other diagnostic axis I whose treatment take precedence over the treatment of OCD (bipolar affective disorder; dependence alcohol; schizophrenia or psychotic disorders; dementia)
* Presence of other neurological diseases or severe clinical as neurodegenerative diseases, severe aphasia, malignancies activity, epilepsy, previous head injury, congestive heart failure or chronic obstructive pulmonary disease stage III or IV;
* Presence of severe suicidal ideation (Structured planning suicide or attempted suicide in the past 4 weeks);
* Pregnancy;
* Inability to provide informed consent;
* Specific contraindication to tDCS: ( metal plates on the head, anatomic changes.);
* In relation to the current use of psychotropic drugs will be permitted, provided they are in doses stable for at least 6 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
change in baseline Yale-Brown Obsessive Compulsive Scale score | weeks 4,6,9,12

SECONDARY OUTCOMES:
Beck Depression Inventory symptoms, | baseline, weeks 6 and 12
Beck Anxiety Inventory | baseline, week 6 and 12
Global Clinical Impression Scale - improvement | baseline, week 6 and 12

CONTACTS AND LOCATIONS:
Locations (1):
- USP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Silva RM, Brunoni AR, Miguel EC, Shavitt RG. Transcranial direct current stimulation for treatment-resistant obsessive-compulsive disorder: report on two cases and proposal for a randomized, sham-controlled trial. Sao Paulo Med J. 2016 Sep-Oct;134(5):446-450. doi: 10.1590/1516-3180.2016.0155010716. PMID 27901245